CLINICAL TRIAL: NCT07295886
Title: Observational Study on the Use of Topical Nifedipine 0.3% and Lidocaine 1.5% in Acute Uncomplicated Hemorrhoidal Disease
Brief Title: Topical Nifedipine 0.3% Plus Lidocaine 1.5% for Uncomplicated Hemorrhoidal Disease
Acronym: NILOS
Status: Recruiting | Type: Observational
Sponsor: Cardarelli Hospital (Other)
Collaborators: Neopharmed Gentili S.p.A. (Industry)
Responsible Party: Principal Investigator, Antonio Brillantino, MD, PhD, Cardarelli Hospital
Other Study IDs: Nilos
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhoid Bleeding; Hemorrhoids Prolapse; Hemorrhoid Pain; Hemorrhoid; Topical Administration
Keywords: nifedipine 0.3% plus lidocaine 1.5%; uncomplicated hemorrhoidal disease; hemorrhoids symptoms
MeSH Terms: conditions — Hemorrhoids | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute, uncomplicated hemorrhoidal disease: 80 patients with acute, uncomplicated hemorrhoidal disease who sign informed consent and meet all eligibility criteria.
  Interventions: Drug: topical nifedipine 0.3% plus lidocaine 1.5%

INTERVENTIONS:
Drug: topical nifedipine 0.3% plus lidocaine 1.5% — Transrectal and perianal application of nifedipine 0.3% plus lidocaine 1.5% cream twice daily for at least 21 days in patients with acute, uncomplicated hemorrhoidal disease

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of topical nifedipine 0.3% plus lidocaine 1.5% for uncomplicated hemorrhoidal disease. The main question it aims to answer is:

Does topical nifedipine 0.3% plus lidocaine 1.5% lower symptoms in patients with uncomplicated acute hemorrhoidal disease? Participants already taking nifedipine 0.3% plus lidocaine 1.5% as part of their regular medical care for hemorrhoidal disease will undergo four visits over a 30-day period, including two telephone contacts and two in-person visits.

DETAILED DESCRIPTION:
Prospective, observational, single-center study involving the administration of topical nifedipine 0.3% plus lidocaine 1.5%, rectally and perianally twice daily for at least 21 days, in patients with uncomplicated hemorrhoidal disease.

The Primary Objective is to evaluate the real-world effectiveness of topical nifedipine 0.3% + lidocaine 1.5% in acute, uncomplicated hemorrhoidal disease, with particular focus on symptom resolution, assessed through the analysis of changes in the HDSS (Hemorrhoidal Disease Symptom Score) questionnaire. The Secondary Objectives include the assessment of topical combinations effect on reduction of hemorrhoidal prolapse (down-staging), its impact on patients' quality of life and its role in preventing hemorrhoidal thrombosis.

Eligible patients-those who meet inclusion/exclusion criteria, sign informed consent, and receive a clinically indicated therapeutic protocol within 5 days of baseline evaluation (dietary recommendations, hydration, and topical therapy)-will undergo 4 assessments over approximately 30 days:

T0: Baseline visit within 5 days of starting nifedipine 0.3% + lidocaine 1.5% T1: Telephone contact at day 10 T2: In-person visit at day 21 T3: Telephone contact at day 30

The study includes an enrollment period of 10 months, an observation period of ~30 days and total duration of ~12 months

Data will be collected at the study center and entered by the investigator or designated personnel into a web-based electronic database (e-CRF), structured according to the study flow-chart.

The study plans to enroll 80 patients. This number is justified by the expected change in HDSS score between baseline (T-1) and T2 (day 21). Assuming a standard deviation of ~5 points, a sample of 70 patients ensures a precision of 1.2 points for 95% confidence intervals. To account for a 10% drop-out rate, the final sample size is set at 80 patients.

Continuous variables will be described using mean ± SD, quartiles (25%, 50%, 75%), and min/max.

Categorical variables using absolute frequencies and percentages. Statistical analysis will be performed using SAS 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-75 years.
* Clinical or anoscopic diagnosis of acute hemorrhoidal disease with prolapse severity between Grade II and IV (Goligher), possibly associated with external congestion.
* Patients who started treatment with nifedipine 0.3% + lidocaine 1.5% within the past 5 days.
* Availability of clinical evaluations at treatment initiation (proctologic visit and HDSS, SHS-HD, VAS scales).
* Ability to understand the informed consent.
* Signed informed consent.

Exclusion Criteria:

* Acute hemorrhoidal disease complicated by thrombosis or strangulation.
* Coagulopathies.
* Active neoplastic disease.
* Treatment with anticoagulants and/or chemotherapeutic agents.
* Hypersensitivity to active substances, especially lidocaine (and other amide-type local anesthetics) or excipients.
* Severe hypotensive states or cardiovascular insufficiency.
* Pregnancy or breastfeeding.
* Participation in clinical trials involving investigational drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 80 patients with acute, uncomplicated hemorrhoidal disease who sign informed consent and meet all eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-05-02 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
Change in HDSS (hemorrhoidal disease symptom score) questionnaire, analyzed using paired t-test or Wilcoxon signed-rank test according to data distribution. The total HDSS ranges from 0 to 20, with higher scores indicating greater symptom severity. | From enrollment to the 30-day follow-up

SECONDARY OUTCOMES:
Quality of life related to hemorrhoidal disease | From baseline to 30 day follow-up
  Change in SHS-HD (Short Health Scale for Hemorrhoidal Diseases score) analyzed using paired t-test or Wilcoxon signed-rank test, depending on data distribution. Total SHS-HD score ranges from 0 to 28, with higher scores indicating greater symptom severity
Hemorroidal Pain | From baseline to 30 day follow-up
  Change in VAS (Visual analogue scale) score (assessed with paired t-test or Wilcoxon test). Total VAS score ranges from 0 to 10 with higher score indicating great symptom severity.
Hemorrhoidal prolapse down-staging | From baseline to 30 day follow-up
  Evaluation of Prolapse down-staging with Cochran-Armitage test for ordinal data. Prolapse grading is evaluated by Goligher scale which ranges from grade I to grade IV, with increasing severity. Particularly, grade 1: Hemorrhoids that bleed but do not prolapse; Grade 2: Hemorrhoids that prolapse but spontaneously reduce; Grade 3: Hemorrhoids that prolapse but have to be manually reduced; Grade 4: Hemorrhoids that prolapse but cannot be reduced

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera "Antonio Cardarelli", Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Result] Brillantino A, Renzi A, Talento P, Brusciano L, Marano L, Grillo M, Maglio MN, Foroni F, Palumbo A, Sotelo MLS, Vicenzo L, Lanza M, Frezza G, Antropoli M, Gambardella C, Monaco L, Ferrante I, Izzo D, Giordano A, Pinto M, Fantini C, Gasparrini M, Schiano Di Visconte M, Milazzo F, Ferreri G, Braini A, Cocozza U, Pezzatini M, Gianfreda V, Di Leo A, Landolfi V, Favetta U, Agradi S, Marino G, Varriale M, Mongardini M, Pagano CEFA, Contul RB, Gallese N, Ucchino G, D'Ambra M, Rizzato R, Sarzo G, Masci B, Da Pozzo F, Ascanelli S, Liguori P, Pezzolla A, Iacobellis F, Boriani E, Cudazzo E, Babic F, Geremia C, Bussotti A, Cicconi M, Sarno AD, Mongardini FM, Brescia A, Lenisa L, Mistrangelo M, Zuin M, Mozzon M, Chiriatti AP, Bottino V, Ferronetti A, Rispoli C, Carbone L, Calabro G, Tirro A, de Vito D, Ioia G, Lamanna GL, Asciore L, Greco E, Bianchi P, D'Oriano G, Stazi A, Antonacci N, Renzo RMD, Poto GE, Ferulano GP, Longo A, Docimo L. The Italian Unitary Society of Colon-Proctology (Societa Italiana Unitaria di Colonproctologia) guidelines for the management of acute and chronic hemorrhoidal disease. Ann Coloproctol. 2024 Aug;40(4):287-320. doi: 10.3393/ac.2023.00871.0124. Epub 2024 Aug 30. PMID 39228195
- [Result] Tarasconi A, Perrone G, Davies J, Coimbra R, Moore E, Azzaroli F, Abongwa H, De Simone B, Gallo G, Rossi G, Abu-Zidan F, Agnoletti V, de'Angelis G, de'Angelis N, Ansaloni L, Baiocchi GL, Carcoforo P, Ceresoli M, Chichom-Mefire A, Di Saverio S, Gaiani F, Giuffrida M, Hecker A, Inaba K, Kelly M, Kirkpatrick A, Kluger Y, Leppaniemi A, Litvin A, Ordonez C, Pattonieri V, Peitzman A, Pikoulis M, Sakakushev B, Sartelli M, Shelat V, Tan E, Testini M, Velmahos G, Wani I, Weber D, Biffl W, Coccolini F, Catena F. Anorectal emergencies: WSES-AAST guidelines. World J Emerg Surg. 2021 Sep 16;16(1):48. doi: 10.1186/s13017-021-00384-x. PMID 34530908
- [Result] Antropoli C, Perrotti P, Rubino M, Martino A, De Stefano G, Migliore G, Antropoli M, Piazza P. Nifedipine for local use in conservative treatment of anal fissures: preliminary results of a multicenter study. Dis Colon Rectum. 1999 Aug;42(8):1011-5. doi: 10.1007/BF02236693. PMID 10458123
- [Result] Perrotti P, Bove A, Antropoli C, Molino D, Antropoli M, Balzano A, De Stefano G, Attena F. Topical nifedipine with lidocaine ointment vs. active control for treatment of chronic anal fissure: results of a prospective, randomized, double-blind study. Dis Colon Rectum. 2002 Nov;45(11):1468-75. doi: 10.1007/s10350-004-6452-1. PMID 12432293
- [Result] Perrotti P, Antropoli C, Molino D, De Stefano G, Antropoli M. Conservative treatment of acute thrombosed external hemorrhoids with topical nifedipine. Dis Colon Rectum. 2001 Mar;44(3):405-9. doi: 10.1007/BF02234741. PMID 11289288
- [Result] Thomson WH. The nature of haemorrhoids. Br J Surg. 1975 Jul;62(7):542-52. doi: 10.1002/bjs.1800620710. PMID 1174785
- [Result] GASS OC, ADAMS J. Hemorrhoids; etiology and pathology. Am J Surg. 1950 Jan;79(1):40-3. doi: 10.1016/0002-9610(50)90189-9. No abstract available. PMID 15399351